CLINICAL TRIAL: NCT00011856
Title: Linkage Analysis of Familial Intracranial Aneurysms
Brief Title: Genetic Analysis of Familial Brain Aneurysms
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010101; 01-HG-0101
Record Dates: First submitted 2001-03-01; First posted 2001-03-02 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-03

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial Aneurysms; Cerebral; Loci; Susceptibility Genes; Cerebral Aneurysm; Familial Cerebral Aneurysm; Genetics
MeSH Terms: conditions — Intracranial Aneurysm

SUMMARY:
This study will investigate cerebral (brain) aneurysms and their possible inheritance patterns in families. It will try to determine how often brain aneurysms occur in families in which more than one member has had an aneurysm and to find the gene or genes that contribute to their development.

People in families in which more than one family member had a cerebral aneurysm are eligible for this 1-day study. They will undergo the following procedures:

* Blood will be drawn (no more than 3 to 4 tablespoons) for research to identify genes that contribute to the development of brain aneurysms.
* A magnetic resonance angiograph (MRA) scan will be done to examine a specific brain area where aneurysms typically occur. Magnetic resonance imaging uses a strong magnetic field and radio waves to produce images of the brain and detect abnormalities.

If a more detailed picture of the brain is needed than can be obtained with MRA, a more specific MRA scan will be done using a contrast dye to enhance the images.

Patients may be invited to participate in related NIH research studies.

DETAILED DESCRIPTION:
This study is designed to explore the genetics of familial cerebral aneurysms. Families in which more than one person has had a known cerebral aneurysm will be studied. Family histories will be obtained and participants identified who are willing to come to the NIH Clinical Center for an MRAngiograph and venipuncture. DNA will be isolated and linkage studies undertaken to identify loci involved in the etiology of familial cerebral aneurysms, using standard linkage approaches.

ELIGIBILITY:
INCLUSION CRITERIA:

Participants and their relatives that are affected or at a higher risk for cerebral aneurysms will be enrolled in this protocol.

EXCLUSION CRITERIA:

For the MR Angiograph portion of the study, any participant that is not able to sign the Clinical Center consent form due to metal implants, pregnancy, claustrophobia, or an allergy to gadolinium as a contrast will be excluded from the imaging part of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2001-02; Study Completion 2002-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States